CLINICAL TRIAL: NCT04289844
Title: Efficacy of a Physiotherapy Intervention Through an Elastic-explosive Strength Training Combined With Active Joint Mobilizations, on the Improvement of the Efficiency of Repeated Vertical Jumping in Basketball Players
Brief Title: Elastic-explosive Strength Training Combined With Active Joint Mobilizations in Basketball Players
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Lockdown
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Jump
Record Dates: First submitted 2020-02-27; First posted 2020-02-28 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Basketball Players
Keywords: Active mobilizations; Strength; Endurance; Vertical Jump; Physiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Each session of the intervention will have a duration of 15 minutes of specific training taking place two sessions a week, during a period of 5 weeks. The exercises will be performed in the first 15 minutes of the training session. The intervention will include specific exercises of elastic-explosive strength and resistance strength
  Interventions: Other: Elastic-explosive and resistance strength
- Control group (Active Comparator): Each session of the intervention will have a duration of 10 minutes of specific training taking place two sessions a week, during a period of 5 weeks. The exercises will be performed in the first 15 minutes of the training session. The intervention will include specific exercises of elastic-explosive strength
  Interventions: Other: Elastic-explosive strength

INTERVENTIONS:
Other: Elastic-explosive and resistance strength — The resistance exercises are: running (3 minutes), 2 farmers carrying marching, 3 side to side ankle hops, 4 plyo lunge jump, 5 lateral jump over barrier, 2 monopodalic jump with ball pass, 3 board throw with half court sprint, 4 lateral shuffle mirror, and 5 combo finisher 4x4.
  Plyometric exercises are: ankle rotations, knee extension, squat, hip flexion-extension, knee and ankle, ankle mobilizations, squat with rise, pelvis ante / retroversion, global mobilization, stride
  Arms: Experimental group
Other: Elastic-explosive strength — Plyometric exercises are: ankle rotations, knee extension, squat, hip flexion-extension, knee and ankle, ankle mobilizations, squat with rise, pelvis ante / retroversion, global mobilization, stride
  Arms: Control group

SUMMARY:
The specific training of the elastic-explosive force of the muscles involved in vertical jump and active mobilizations is used to improve the quality of the jump. It is also intended to reduce the loss of centimeters, recovery times and fatigue produced during a series of vertical jumps.

The objective of the study is to assess the effectiveness of active mobilizations together with specific training in lower limbs, in ankle mobility, the perception of effort and the height and resistance of vertical jumping in amateur basketball players.

Randomized clinical study. 50 basketball players from 20 to 35 years will be randomized to the study groups: control group (resistance strength exercises, elastic-explosive force) and experimental group (resistance strength exercises, elastic-explosive force together with active mobilizations). The dependent variables will be: repeated jump (15 second Jump test, my Jump 2), maximum vertical jump (CMJ free arms, my Jump 2), subjective perception of effort (Borg scale) and ankle dorsiflexion (goniometer). The sample distribution will be calculated using a Kolmogorov-Smmirnof analysis. The changes after each evaluation will be analyzed with the t-student test and with an ANOVA of repeated measures the intra and intersubject effect will be observed. The effect size will be calculated using Cohen's formula.

It is expected to observe an improvement in the resistance of vertical jumps, with a decrease in the loss of centimeters in the repetitions of jumps.

ELIGIBILITY:
Inclusion Criteria:

* Basketball players in the Community of Madrid
* Male
* With an age range of 18 to 35 years
* Federated

Exclusion Criteria:

* Athletes who present an injury at the time of the study
* Who are receiving some parallel physiotherapy intervention
* Have an injury during the experimental or follow-up phase
* Have not signed the informed consent document

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline maximum vertical jump after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The My Jump 2 application will be used. With the video we can see the moment when the feet do not touch the ground and with this data the application automatically calculates the height in centimeters. From a squat position, the player will have to perform a vertical jump, landing in the same starting position.

SECONDARY OUTCOMES:
Change from baseline resistance of the explosive force after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The 15 sec repeated jump test will assess the resistance of the explosive force. With the My Jump 2 application we will calculate the height in repeated jumps in 15 seconds. To do this, we will ask the athlete to, from a squat position, perform 15 repeated vertical jumps, returning to the starting position every time.
Change from baseline subjective perception of effort after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  We will use the modified Borg scale with a scoring range of 1 to 10 points (the higher the score, the greater the perception of effort). The concept of perceived effort is a subjective assessment that indicates the person's opinion regarding the intensity of the work performed. 1 indicates little fatigue, 10 is the maximum effort perceived by the athlete
Change from baseline dorsal ankle flexion after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  This variable will be measured with the use of a goniometer. With the athlete standing, from a stride position, with the first finger placed 10 cm from the wall, we will ask him to do a knee flexion towards the wall, with the heel always resting on the floor. We will place the goniometer axis in the center of the outer malleolus. The fixed arm will be parallel to the ground, while the mobile arm will be aligning the fibula. The unit of measure is the degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain